CLINICAL TRIAL: NCT00987012
Title: The Influence of Fortified Pomegranate Juice (Punica Granatum) on Seasonal Influenza and Swine Flu Patients - A Prospective Randomized Trial
Brief Title: The Influence of Fortified Pomegranate Juice (Punica Granatum) on Seasonal Influenza and Swine Flu Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Gan shmuel Group (Other)
Responsible Party: Dr. Gershon Keren, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0044-09-HYMC
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Influenza A; Swine Flu
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pomegranate juice (Experimental)
  Interventions: Dietary Supplement: Pomegranate juice
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Pomegranate juice — Twice daily ingestion of pomegranate juice over 4-5 days
  Arms: Pomegranate juice
Dietary Supplement: Placebo drink — Twice daily ingestion of placebo drink over 4-5 days
  Arms: Placebo drink

SUMMARY:
It has been shown in laboratory studies that pomegranate juice contains anti-viral action against influenza. The researchers wish to investigate the effect of pomegranate juice on patients suffering from influenza A (seasonal or swine flu).

ELIGIBILITY:
Inclusion Criteria:

* Individuals confirmed and suffering from Influenza A

Exclusion Criteria:

* Individuals suffering from influenza included in the high risk group

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Early relief of influenza symptoms | Within one week

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel